CLINICAL TRIAL: NCT04054739
Title: Effects of Robotic Gait Training on Cortical Activity and Gait Function in Hemiparetic Stroke
Brief Title: Cortical Activity and Gait Function for Robotic Gait Training in Hemiparetic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Rehabilitation Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Joon-Ho Shin, Team manager, National Rehabilitation Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRC-2017-02-015
Record Dates: First submitted 2019-08-12; First posted 2019-08-13 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Stroke
Keywords: robot-assisted gait training; cortical activity; gait kinematics; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted gait training (Experimental): experimental group that applied the end-effector robot-assisted gait training
  Interventions: Device: Robot-assisted gait training
- Treadmill gait training (Active Comparator): control group that applied the treadmill gait training
  Interventions: Device: Treadmill gait training

INTERVENTIONS:
Device: Robot-assisted gait training — intervention with robot-assisted gait training
  Arms: Robot-assisted gait training
Device: Treadmill gait training — intervention with treadmill gait training
  Arms: Treadmill gait training

SUMMARY:
Effects of robot-assisted gait training on cortical activity and gait function in hemiparetic stroke

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegic patients secondary to first cerebrovascular accidents
* Functional ambulation category score 3
* 3 months ≤ Onset ≤ 12 months
* Korean Mini-Mental State Examination score > 24

Exclusion Criteria:

* History of surgery of affected lower limb
* Fracture of affected lower limb

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
oxygenated hemoglobin levels | 4 weeks from baseline
  cortical activity of primary sensorimotor cortex, premotor cortex, supplementary motor areas, pre-supplementary motor areas, prefrontal cortex during gait
Range of motion of ankle, knee, and hip joint | 4 weeks from baseline
  ankle, knee, and hip joint motion of sagittal plane during gait

SECONDARY OUTCOMES:
oxygenated hemoglobin levels | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  cortical activity of primary sensorimotor cortex, premotor cortex, supplementary motor areas, pre-supplementary motor areas, prefrontal cortex during gait
Range of motion of ankle, knee, and hip joint | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  ankle, knee, and hip joint motion of sagittal plane during gait
Berg Balance Scale | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Berg Balance Scale assess the functional balance ability of participants with observation of 14 tasks, representing functional movements common in daily life. Each task is scored on a five-point scale (0-4) following the guidelines of the test developers, and the maximum score on this test is 56 which indicates balance ability within the normal range.
Fugl-Meyer Assessment | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Fugl-Meyer Assessment uses to examine the motor function and coordination of affected lower extremity. It includes 17 items of a 3-point ordinal scale, ranging 0-34, with higher scores indicating lower impairment.
10m walk test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  10m walk test is used to examine gait speed, in which participant was asked to walk on a 14 meter of walkway wearing harness with two conditions; with the fastest speed or with self-selected comfortable speed.
Functional ambulation category | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Functional Ambulation Category is used to assess gait ability with 6 levels ranging from 0 to 5 on the basis of the amount of physical support required, regardless of use of an assistive device
Falls efficacy scale | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Korean version of Falls efficacy scale asks subjects to rank their confidence about their ability not to fall while performing a variety of activities of daily living with a maximum score of 100
Beck depression inventory | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  21-question multiple-choice self-report inventory, one of the most widely used psychometric tests
Stroke impact scale | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  health-related quality of life poststroke across 8 domains using a 5-point Likert scale, with the score ranging from 0 to 100 and a higher score indicating better health status
Dynamic gait index | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  a clinical tool to assess gait, balance and fall risk
Timed up and go test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  a simple test used to assess a person's mobility and requires both static and dynamic balance
modified Barthel index | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Measure of physical disability used widely to assess behaviour relating to activities of daily living for stroke patients
dual task - COWAT | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Controlled Oral Word Association Test, abbreviated COWA or COWAT, is a verbal fluency test that measures spontaneous production of words belonging to the same category or beginning with some designated letter.
dual task - digit span test | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  The digit span test is a way of measuring the storage capacity of a person's working memory.
Electromyography of lower extremities | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Muscle activity of tibialis anterior, medial gastrocnemius, vastus medialis, biceps femoris, gluteus medius during gait.
Plantar pressure | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Plantar pressure (great toe, little toe, medial meta, lateral meta, medial arch, lateral arch, heel) during gait
Spatiotemporal gait parameter data | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  step length, step time, swing time, double limb support time during gait
deoxygenated hemoglobin levels | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  cortical activity of primary sensorimotor cortex, premotor cortex, supplementary motor areas, pre-supplementary motor areas, prefrontal cortex during gait
total hemoglobin levels | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  cortical activity of primary sensorimotor cortex, premotor cortex, supplementary motor areas, pre-supplementary motor areas, prefrontal cortex during gait
Balance test using force plate | baseline, 2 weeks after baseline, 4 weeks after baseline, 8 weeks after baseline
  Static standing balance as measured using a force plate: Changes in center-of-pressure velocity and area

CONTACTS AND LOCATIONS:
Overall Officials: Joon-Ho Shin, MS, Principal Investigator — National Rehabilitation Center
Locations (1):
- National Rehabilitation Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim H, Park G, Shin JH, You JH. Neuroplastic effects of end-effector robotic gait training for hemiparetic stroke: a randomised controlled trial. Sci Rep. 2020 Jul 27;10(1):12461. doi: 10.1038/s41598-020-69367-3. PMID 32719420